CLINICAL TRIAL: NCT01680679
Title: Influenza Immunization of Children in India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: All India Institute of Medical Sciences (Other); International Clinical Epidemiology Network (INCLEN) TRUST (Network); University of Alabama at Birmingham (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13-0210; U01IP000475 (NIH)
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Influenza
Keywords: Influenza; India; Children; Trivalent Influenza Vaccine (TIV); Inactivated poliovirus vaccine (IPV); Direct influenza vaccine effectiveness; Total influenza vaccine effectiveness; Indirect influenza vaccine effectiveness
MeSH Terms: conditions — Influenza, Human | interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Inactivated Trivalent Influenza Vaccine (Experimental): Inactivated trivalent influenza vaccine (TIV), split virion
  Interventions: Biological: Inactivated Trivalent Influenza Vaccine (TIV)
- Inactivated Polio Vaccine (Placebo Comparator): Inactivated poliovirus vaccine (IPV), trivalent
  Interventions: Biological: Inactivated poliovirus vaccine (IPV), trivalent
- Surveillance arm (No Intervention): Those ineligible for vaccination will be enrolled for febrile acute respiratory illness (FARI) surveillance to assess indirect effects of vaccination in household members.

INTERVENTIONS:
Biological: Inactivated Trivalent Influenza Vaccine (TIV)
  Arms: Inactivated Trivalent Influenza Vaccine
Biological: Inactivated poliovirus vaccine (IPV), trivalent
  Arms: Inactivated Polio Vaccine

SUMMARY:
Influenza viruses are significant causes of human illness and death in developed and developing countries. This study will measure the ability of influenza vaccine given to children in India to protect both the children and unimmunized persons around them from influenza. It will also determine whether the best time to immunize in a country like India that has both summer and winter outbreaks of influenza is in the fall, as is done now, or whether immunization should be in the spring to protect against influenza infections in the summer.

DETAILED DESCRIPTION:
Although influenza vaccines are used routinely in the United States, including in young children, influenza vaccines have not seen widespread use in India. This is likely contributed to by the lack of information from India about disease burden due to influenza and because influenza vaccines have not been tested for efficacy in India. In addition, because young children are thought to be important in the spread of influenza in families, it is possible immunization of children against influenza will reduce influenza infections among older children and adults in the home. The study described here is an extension of an earlier study (ClinicalTrials.gov NCT00934245) that tested the use of immunization against influenza in the fall. The current study will administer influenza vaccine in the spring prior to the summer monsoon rains that are associated with peaks of influenza activity in parts of India. Reduction of influenza infections among the influenza immunized children and their household members will be compared to the children and household members in the control vaccine group.

ELIGIBILITY:
Inclusion Criteria:

Inclusion in either vaccine group (TIV or IPV) will require ages 6 months through 10 years of age.

All individuals in enrolled households will be eligible for enrollment into surveillance arm.

Exclusion Criteria:

Exclusion criteria from the vaccine groups includes known allergy to eggs, or hypersensitivity to other components of the vaccines.

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18163 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Laboratory-confirmed influenza infection in vaccinated child | 1 year

SECONDARY OUTCOMES:
Laboratory-confirmed influenza infection in household member of a vaccinated child. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Sullender, MD, Principal Investigator — University of Colorado, Denver; Shobha Broor, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- Comprehensive Rural Health Services Project, Ballabgarh, Haryana, India